CLINICAL TRIAL: NCT04585867
Title: Liposomal Bupivacaine vs Bupivacaine for Pain Control After Sternotomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jared Staab, DO, Study Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00140472
Record Dates: First submitted 2020-09-24; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Pain Management; Sternotomy
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal bupivacaine (Active Comparator): Exparel (266mg) given by surgeon just prior to sternal closure
  Interventions: Drug: Exparel
- Bupivacaine (Active Comparator): 40ml of 0.125% bupivacaine given by surgeon just prior to sternal closure
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Exparel — The injections will be performed under direct guidance by the cardiac surgeon at bilateral sternal-costal interspaces 1.5 cm lateral the sternal boarder at levels 2-6 in divided doses (2 ml/injection) just before the closure of the sternum near the end of the surgical procedure. The final 20 ml will be injected into the skin incision after closure
  Arms: Liposomal bupivacaine
Drug: Bupivacaine — The injections will be performed under direct guidance by the cardiac surgeon at bilateral sternal-costal interspaces 1.5 cm lateral the sternal boarder at levels 2-6 in divided doses (2 ml/injection) just before the closure of the sternum near the end of the surgical procedure. The final 20 ml will be injected into the skin incision after closure
  Arms: Bupivacaine

SUMMARY:
Researchers hope to learn whether giving the longer-acting local anesthetic liposomal bupivacaine prior to closing the sternum is more effective in managing pain following sternotomy, than in patients who received standard bupivacaine before sternal closure. Researchers will measure this based on how much IV pain medication is used, rates on confusion, and time to remove the breathing tube.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 who present for elective open heart surgery that requires a sternotomy.

Exclusion Criteria:

* Urgent and emergency procedures,
* preexisting sternal infections,
* prior sternotomy,
* preexisting pain syndromes,
* current chronic home opioid use,
* anterior rib or sternal masses,
* allergy to any of the components of liposomal bupivacaine and plain bupivacaine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption in morphine equivalents | 0 hours post-surgery
  Opioid consumption in morphine equivalents
Opioid consumption in morphine equivalents | 12 hours post-surgery
  Opioid consumption in morphine equivalents
Opioid consumption in morphine equivalents | 24 hours post-surgery
  Opioid consumption in morphine equivalents
Opioid consumption in morphine equivalents | 36 hours post-surgery
  Opioid consumption in morphine equivalents
Opioid consumption in morphine equivalents | 48 hours post-surgery
  Opioid consumption in morphine equivalents
Opioid consumption in morphine equivalents | 60 hours post-surgery
  Opioid consumption in morphine equivalents
Opioid consumption in morphine equivalents | 72 hours post-surgery
  Opioid consumption in morphine equivalents

SECONDARY OUTCOMES:
Time to extubation in minutes will be retrieved via the electronic medical record | 30 days post operative
  Time to extubation in minutes will be retrieved via the electronic medical record
Presence of sternal wound infection | 4-6 weeks postoperative visit
  Presence of sternal wound infection will be retrieved via electronic medical record and at 30 day follow up for Society of Thoracic Surgery (STS) database data as well as sternal infection documented at standard postoperative visit at 4-6 weeks
Postoperative delirium as assessed by Confusion Assessment Method (CAM)-ICU | 30 days post operative
  Postoperative delirium as assessed by CAM-ICU at hours 0,12,24,36,48,60,and 72 hours post-surgery will be retrieved via the electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Jared Staab, DO, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States